CLINICAL TRIAL: NCT06671964
Title: The Impact of School-Based Intervention for 9-13-year-old School Children with Overweight and Obesity: Nutrition Knowledge, Attitudes, Self-Efficacy, Fruit and Vegetable Intake, and Anthropometry
Brief Title: The Impact of School-Based Intervention for 9-13-year-old School Children with Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Sara Zuarub, Principal Investigator, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERSC_2022_744
Record Dates: First submitted 2024-08-29; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Overweight Children; Obese Children and Adolescents
Keywords: Overnutrition; Nutrition Disorders; Body Weight; Overweight; SchoolChildren; peer pressure
MeSH Terms: conditions — Overnutrition; Nutrition Disorders; Body Weight; Overweight | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: 1. Educational sessions
  2. Anthropometric measurements
  3. Questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- students one-one (Other): 1. During the intervention, 30-minute in person sessions and lectures are held on a one-on-one basis .
  2. Lectures were conducted daily for five days during the first month of the intervention
  3. The students were exposed to the school nutrition education curriculum, which may also be considered an intervention as it introduced students to new nutrition knowledge. The school nutrition education curriculum presented general information about nutrition in accordance with official guidelines issued by the UAE Ministry of Education. Topics covered included the dangers of obesity, the prevalence of obesity in the UAE, and potentially effective ways to prevent this problem, the information in this program was broad and did not provide practical recommendations to students except for a set of general suggestions.
  4. The topics covered included a healthy eating lifestyle, energy balance, food portion control, healthy snacking, the importance of physical activity and healthy eating, dietary
  Interventions: Other: Anthropometric measurements; Other: Questionnaire; Other: Educational sessions
- Peers (Other): 1. 30-minute in person sessions were introduced to all the school children, and 10-minute question-and-answer sections were held at the end of each lesson to support knowledge acquisition.
  2. Lectures were conducted daily for five days in the first month of the study.
  3. The students were exposed to the school nutrition education curriculum, which may also be considered an intervention as it introduced students to new nutrition knowledge. The school nutrition education curriculum presented general information about nutrition in accordance with official guidelines issued by the UAE Ministry of Education. Topics covered included the dangers of obesity, the prevalence of obesity in the UAE, and potentially effective ways to prevent this problem, the information in this program was broad and did not provide practical recommendations to students except for a set of general suggestions.
  4. The topics covered included a healthy eating lifestyle,
  Interventions: Other: Educational sessions
- Control group (No Intervention): The students in the control group did not receive any nutrition intervention except for the usual school curriculum-based nutrition education program. Participants in the intervention and control groups were recruited from different sections of the same schools.
- parents (Other): 1. 30-minute in person sessions and 10-minute question-and-answer sections were held at the end of each lesson to support knowledge acquisition.
  2. Lectures were conducted daily for five days in the first month of the study.
  Interventions: Other: Educational sessions

INTERVENTIONS:
Other: Anthropometric measurements — Anthropometric measurements of the students, including weight, height, muscle mass, fat quantity, and waist circumference, were measured. The WHO BMI charts were utilized for classification. Stratified Random selection
  Arms: students one-one
Other: Questionnaire — The collection of data was performed using the "Atlas questionnaire" (Al-Hazzaa et al., 2011) and "nutrition knowledge and healthy lifestyle behavior" questionnaire (Kalender et al., 2011) with additional questions related to self-efficacy and dietary practices adapted from the literature (Becher, 2009; Voss et al., 2017; Kowalski et al., 2004). Stratified Random selection
  Arms: students one-one
Other: Educational sessions — The topics that covered included a healthy eating lifestyle, energy balance, food portion control, healthy snacking, the importance of physical activity and healthy eating, dietary practices, and nutrition-related self-efficacy.
  Arms: Peers; parents; students one-one

SUMMARY:
Childhood obesity is a major issue for the United Arab Emirates (UAE). Interventions modifying people's nutritional behavior and changing their dietary habits can potentially address this problem. This study assessed the effectiveness of the 6-month school-based nutritional educational intervention on fruit and vegetable intake, nutrition knowledge, anthropometric measures, and practice, attitude, and self-efficacy measures.

DETAILED DESCRIPTION:
The problem of childhood obesity is a critical issue for the UAE. Findings of recent studies illustrate that nutritional interventions seeking to modify people's nutritional behavior and change their dietary habits have the potential to address this problem. This article reports the results of the study that was dedicated to the influence of the school-based nutritional educational intervention on fruit and vegetable intake, anthropometric measures, practice, attitude, self-efficacy, and knowledge scores of schoolchildren. The intervention was carried out among 9-13-year-old schoolchildren at public schools from Dubai and Sharjah (n=403). The sample included three groups, including the control group (n=114), Intervention Group 1 (n=148), and Intervention Group 2 (n=141). The control group was exposed to a conventional curriculum on healthy nutrition. Group 1 participated in the intervention involving children, and Group 2 participated in the intervention involving students, peers, and parents.

ELIGIBILITY:
Inclusion Criteria:

* WHO BMI-for-age growth charts, Students with BMI from the 85th to the 95th percentile were categorized as "overweight," and those who were above the 95th percentile were categorized as "obese"
* Attending Government school.
* Within Grades 6-9.
* Live in Dubai or Sharjah
* Female and male students

Exclusion Criteria:

* Students with BMI below the 85th percentile for the WHO BMI-for-age growth charts.
* Not attending a government school
* Living in another emirate (not Dubai or Sharjah)

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 403 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Nutrition Knowledge and Self-Efficacy | 6 months
  - Change in students' knowledge and self-efficacy scores from baseline values in overweight and obese UAE students aged 9-13 using a validated questionnaire(Arab Teens Lifestyle Questionnaire).
  The statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) software, and the IBM, USA computer software (version 29).
  Likert scales, were expressed as weighted mean ± SD. An independent t-test (parametric test) was used to analyze the effect of 2-level qualitative variables on quantitative variables, and one way ANOVA (parametric test) was used to analyze the effect of >2-level qualitative variables on quantitative variables in each questionnaire section
Nutrition Knowledge and Self-Efficacy | 6 months
  - Change in the percentage of children consuming at least five servings of fruits and vegetables and using a validated questionnaire(Arab Teens Lifestyle Questionnaire).
  The statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) software, and the IBM, USA computer software (version 29).
  Likert scales, were expressed as weighted mean ± SD. An independent t-test (parametric test) was used to analyze the effect of 2-level qualitative variables on quantitative variables, and one way ANOVA (parametric test) was used to analyze the effect of >2-level qualitative variables on quantitative variables in each questionnaire section

SECONDARY OUTCOMES:
Anthropometric Data | 6 months
  Change in body measurements(Weight in kilogram, BMI in kg/m^2) The statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) software, and the IBM, USA computer software (version 29).The anthropometric measurements of the control and intervention groups were compared using ANOVA before and after the nutritional education intervention.
Anthropometric Data | 6 months
  Change in body measurements(waist circumference in cm) The statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) software, and the IBM, USA computer software (version 29).The anthropometric measurements of the control and intervention groups were compared using ANOVA before and after the nutritional education intervention.
Anthropometric Data | 6 months
  Change in body measurements( Muscle Mass in kilogram) The statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) software, and the IBM, USA computer software (version 29).The anthropometric measurements of the control and intervention groups were compared using ANOVA before and after the nutritional education intervention.
Anthropometric Data | 6 months
  Change in body measurements( Body Fat percentage using using Tanita BC730W) The statistical analyses were performed using the Statistical Package for the Social Sciences (SPSS) software, and the IBM, USA computer software (version 29).The anthropometric measurements of the control and intervention groups were compared using ANOVA before and after the nutritional education intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Habiba Ali, Study Director — UAEU; ESE Research Office, Study Chair — Emarites School Establishment
Locations (1):
- United Arab Emarites University, Al Ain City, Ain, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwalla N, Chehade L, O'Neill LM, Kharroubi S, Kassis A, Cheikh Ismail L, Al Dhaheri AS, Ali HI, Ibrahim S, Chokor FAZ, Mohamad MN, Ayesh W, Nasreddine L, Naja F. Total Usual Nutrient Intakes and Nutritional Status of United Arab Emirates Children (4 Years-12.9 Years): Findings from the Kids Nutrition and Health Survey (KNHS) 2021. Nutrients. 2023 Jan 2;15(1):234. doi: 10.3390/nu15010234. PMID 36615891